CLINICAL TRIAL: NCT02199652
Title: Reducing Suicidal Ideation Through Treatment of Nightmares-PTSD
Brief Title: Reducing Suicidal Ideation Through Treatment of Nightmares-Post Traumatic Stress Disorder (PTSD)
Acronym: REST-ON PTSD
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Augusta University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 00001365
Record Dates: First submitted 2014-07-18; First posted 2014-07-24 (Estimated); Results first posted 2018-08-21 (Actual); Last update posted 2018-09-18 (Actual); Status verified 2018-08

CONDITIONS: Post Traumatic Stress Disorder; Suicidal Ideation; Nightmares
MeSH Terms: conditions — Stress Disorders, Post-Traumatic; Suicidal Ideation | interventions — Prazosin

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- placebo (Placebo Comparator): placebo pill
  Interventions: Drug: Placebo
- prazosin (Experimental): prazosin pill
  Interventions: Drug: Prazosin

INTERVENTIONS:
Drug: Prazosin
  Arms: prazosin
Drug: Placebo
  Arms: placebo

SUMMARY:
Patients with PTSD, and frequent nightmares, and mild-moderate suicidal ideation, who are already taking a Selective Serotonin Reuptake Inhibitor (SSRI) or Serotonin Norepinephrine Reuptake Inhibitor (SNRI) will be randomized to either prazosin or placebo. The investigators hypothesize that patients receiving prazosin will have a greater reduction in suicidal ideation.

ELIGIBILITY:
Inclusion Criteria:

* PTSD
* Frequent nightmares
* Suicidality

Exclusion Criteria:

* Schizophrenia
* Bipolar
* Substance abuse

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2014-03 (Actual); Primary Completion 2017-09-01 (Actual); Study Completion 2017-12-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: William V McCall, MD, MS, Principal Investigator — Augusta University
Locations (1):
- Georgia Regents University, Augusta, Georgia, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- Placebo: placebo pill
  Placebo
- Prazosin: prazosin pill
  Prazosin
Period: Overall Study
Arm/Group | Placebo | Prazosin
Started | 10 | 10
Completed | 3 | 3
Not Completed | 7 | 7

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo | Prazosin | Total
Number analyzed (Participants) | 10 | 10 | 20
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 10 | 10 | 20
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 43.2 (12.7) | 36.3 (15.9) | 39.8 (14.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 8 | 9 | 17
  Male | 2 | 1 | 3
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 4 | 2 | 6
  White | 6 | 8 | 14
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 10 | 10 | 20

OUTCOME MEASURES:

1. Primary Outcome: Change Score for Scale for Suicide Ideation
Description: There will be data on the Scale for Suicide Ideation collected at the end of each week of treatment up to 8 weeks. Our apriori primary outcome is the change score in Scale for Suicide Ideation from baseline to the last observation.
  This is a self report scale, with 19 items which measure present suicidality, each scored 0-2.
  The total scale has a range from 0-38, with higher scores being worse
Time Frame: change score from baseline to last observation, up to 8 weeks
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Placebo | Prazosin
Number analyzed (Participants) | 10 | 10
units on a scale | 7.6 (1.8) | 8.2 (1.9)

2. Secondary Outcome: Disturbing Dreams and Nightmare Severity Index
Description: This is a self report scale, with 5 items, producing a total score with a range from 0-37. Higher scores are worse. A score greater than 10 is considered to indicate a clinically relevant problem with nightmares and/or bad dreams
Time Frame: 8 weeks
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Placebo | Prazosin
Number analyzed (Participants) | 10 | 10
units on a scale | 9.75 (1.7) | 15.8 (1.8)

3. Secondary Outcome: Insomnia Severity Index
Description: This is a self report scale, with 7 items scored 0-4, producing a total score range 0-28.
  Higher scores are worse Score 0-7 is interpreted as "no insomnia problem" 8-14 "subclinical insomnia" 15-21 "moderate insomnia" 22-28 "severe insomnia"
Time Frame: 8 weeks
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Placebo | Prazosin
Number analyzed (Participants) | 10 | 10
units on a scale | 10.7 (1.2) | 15.4 (1.2)

ADVERSE EVENTS:
Time Frame: 8 weeks
Arm/Group | Placebo | Prazosin
All-Cause Mortality (participants affected / at risk) | 0/10 | 0/10
Serious Adverse Events (participants affected / at risk) | 1/10 | 1/10
Other Adverse Events (participants affected / at risk) | 1/10 | 2/10
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo (N=10) | Prazosin (N=10)
psychiatric hospitalization (Psychiatric disorders) | 1 (1) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo (N=10) | Prazosin (N=10)
fainting (Vascular disorders) | 1 (1) | 2 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2015-04-06): https://cdn.clinicaltrials.gov/large-docs/52/NCT02199652/Prot_SAP_000.pdf